CLINICAL TRIAL: NCT02910765
Title: Methylene Blue and Ozone in Early Sepsis , a Randomized Double Blind Trial
Brief Title: Methylene Blue and Ozone in Early Sepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00009906
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Methylene Blue; Ozone; Oxygen

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M methylene blue and ozone (Active Comparator): intravenous methylene blue and blood mixed with ozone ozone injection in early sepsis patients
  Interventions: Drug: methylene blue; Drug: ozone
- P Placebo (Placebo Comparator): saline and oxygen mixed blood injection in early sepsis patients
  Interventions: Other: saline infusion; Other: oxygen

INTERVENTIONS:
Drug: methylene blue
  Arms: M methylene blue and ozone
Drug: ozone
  Arms: M methylene blue and ozone
Other: saline infusion
  Arms: P Placebo
Other: oxygen
  Arms: P Placebo

SUMMARY:
effects of methylene blue and ozone O3 therapy effects in early sepsis management , and their implications upon outcome

DETAILED DESCRIPTION:
effects of methylene blue on inducible nitric oxide messenger RNA transcription and protein expression are well evident in vasoplegia ,and septic shock . In the same time , ozone O3 therapy is also valuable in immune-modulation in multiple pathologies . our study collaborate both methylene blue and Ozone in early sepsis management , and we will evaluate the global medical progress , ICU stay , Morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* early sepsis Adults patients

Exclusion Criteria:

* cardiac problems Glucose-6-Phosphate-Dehydrogenase Insufficiency Ozone Allergy Recent Myocardial Infarction Active Hyperthyroidism Thrombocytopenia Pregnancy Contraindications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
APACHE score | 7 days

SECONDARY OUTCOMES:
ICU stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Emad Zarief K Said, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No